CLINICAL TRIAL: NCT02112630
Title: Prospective, Single-Center, Open Label, Pilot Study of Safety and Efficacy of Triple Anti-Viral Therapy With Pegylated Interferon, Ribavirin, and Boceprevir in Patients With Genotype 1 Chronic HCV With End Stage Renal Disease
Brief Title: Boceprevir in End Stage Renal Disease (ESRD)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Columbia University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAL5200
Record Dates: First submitted 2014-04-02; First posted 2014-04-14 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C Infection; End Stage Renal Disease
Keywords: Hepatitis C Infection; HCV, genotype 1; End Stage Renal Disease; ESRD; Boceprevir; Pegylated Interferon; Ribavirin
MeSH Terms: conditions — Hepatitis C; Kidney Failure, Chronic | interventions — peginterferon alfa-2a; Ribavirin; N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 - Response Guided Therapy (Experimental): Treatment naive and documented relapsers : Subjects who have never been previously treated with P-IFN +/- ribavirin therapy and those who have documented relapse after P-IFN +/- ribavirin therapy.
  Subjects in group 1 will receive P-IFN alfa 2a or P-IFN alfa 2b and ribavirin for a 4 week lead-in followed by the addition of boceprevir. Based on the patient's HCV-RNA levels at Treatment Week (TW) 8, TW12 and TW24 treatment with be continued for a total duration of 28 to 48 weeks.Subjects will be followed through treatment and up to 24 weeks post treatment.
  Interventions: Drug: P-IFN alfa 2a; Drug: P-IFN alfa 2b; Drug: Ribavirin; Drug: Boceprevir
- Group 2 - Fixed Duration Therapy (Experimental): Partial/Null Responders /Undefined Previous Response, Compensated cirrhosis: Subjects who have compensated cirrhosis, and/or were previously treated with P-IFN +/- ribavirin without SVR (including partial responders, null responders, and those previously treated without adequate documentation of response).
  Subjects in Group 2 will all be assigned to fixed duration therapy.Patients will be treated with P-IFN alfa 2a or P-IFN alfa 2b and ribavirin for a 4 week lead-in followed by the addition of boceprevir for a total of 48 weeks of therapy. Subjects will be followed through treatment and up to 24 weeks post treatment.
  Interventions: Drug: P-IFN alfa 2a; Drug: P-IFN alfa 2b; Drug: Ribavirin; Drug: Boceprevir

INTERVENTIONS:
Drug: P-IFN alfa 2a — P-IFN alfa 2b 0.75 mcg/kg/week
  Other Names: Pegylated-interferon alfa 2a
Drug: P-IFN alfa 2b — P-IFN alfa 2a 135 mcg/kg/week
  Other Names: Pegylated-interferon alfa 2b
Drug: Ribavirin — 200 mg PO once daily or 200 mg PO three times a week
  Other Names: Copegus®
Drug: Boceprevir — 800 mg PO three times daily starting at week 4
  Other Names: Victrelis

SUMMARY:
The purpose of the study is to assess the safety and efficacy of triple therapy with pegylated interferon (P-IFN), ribavirin and boceprevir in patients with genotype 1 chronic Hepatitis C Virus (HCV) infection and end stage renal disease (ESRD) on hemodialysis (HD).

DETAILED DESCRIPTION:
Hepatitis C (HCV) remains the most common chronic infection in the United States with about 3 million people chronically infected. The majority of these patients in the U.S. have genotype 1 HCV infection, which has been the most difficult genotype to treat with the traditional regimen of pegylated-interferon (P-IFN) and ribavirin, leading to sustained virologic response (SVR) in less than 50% of cases. HCV is also an established risk factor for chronic kidney disease (CKD) and end-stage renal disease (ESRD) and unfortunately the treatment is even less successful in these patients mainly limited by increased medication toxicity.

In spring of 2011, the FDA approved two new direct acting antivirals (DAA) for the treatment of chronic genotype 1 HCV, boceprevir and telaprevir, to be used in combination with Peg-IFN and ribavirin. This 'triple therapy' approach has significantly increased the response rate (increased SVR rates to about 80% in those patients who had never been previously treated) representing a significant advance in the field. In addition, several response-guided therapy approaches were tested to determine if treatment duration could be shortened based upon the virologic response on treatment.

To date, there have been no studies evaluating the safety and efficacy of triple therapy in patients with ESRD. However, a single dose pharmacokinetic study of boceprevir in subjects with ESRD on hemodialysis demonstrated that the mean maximum concentration achieved by boceprevir (Cmax) and bioavailability (AUC) were comparable in patients with ESRD and in healthy subjects. Mean t½, median Tmax and mean apparent oral total clearance (CL/F) values were also similar in healthy subjects and patients with ESRD. Boceprevir exposure was also similar on dialysis and non-dialysis days. These data suggest that boceprevir does not need to be adjusted in patients with ESRD on dialysis, and that it is not removed by hemodialysis. To date, there are no studies of telaprevir in ESRD patients.

The investigators therefore aim to study the safety and efficacy of triple therapy using boceprevir in combination with P-IFN and ribavirin in patients with stage 5 CKD (defined as glomerular filtration rate (GFR) < 15 mL.min.1.73m2 on permanent hemodialysis for stage 5). In addition, given the significant toxicity of treatment in this particular patient population, the investigators aim to study the efficacy of response guided therapy in those patients who are eligible for response-guided therapy based on prior studies (treatment naïve patients, and well documented history of relapse with prior treatment with P-IFN and ribavirin).

ELIGIBILITY:
Inclusion Criteria:

1. Adult (ages 18-75)
2. Hepatitis C Virus ribonucleic acid (HCV RNA) 1000 IU/mL or greater
3. Hepatitis C Virus (HCV) genotype 1
4. End stage renal disease on hemodialysis
5. Females of child bearing potential must be using an adequate method of contraception throughout the study and must have a negative pregnancy test prior to the start of treatment.

Exclusion Criteria:

1. Intolerance to peg-IFN or ribavirin with prior treatment course.
2. Prior treatment with protease inhibitor (telaprevir or boceprevir) or experimental protease inhibitor
3. Significant cytopenias:

   1. Absolute neutrophil count (ANC) < 1000/mm3, OR
   2. Hemoglobin (Hgb) <10.5 g/dL, or
   3. Platelet count < 50,000/mm3
4. Significant laboratory abnormalities

   1. Direct bilirubin > 1.5 x upper limit of normal (ULN)
   2. Total bilirubin > 1.6 mg/dL unless due to Gilbert's disease
   3. Prothrombin time (PT)/Partial thromboplastin time (PTT) > 10% above laboratory reference range
   4. Thyroid Stimulating Hormone (TSH) > 1.2 x ULN or < 0.8 x lower limit of normal (LLN)
5. Uncontrolled depression or psychiatric disease
6. Uncontrolled cardiopulmonary or cardiovascular disease
7. Autoimmune diseases except for treated thyroid disease
8. Active substance abuse within 6 months of initiation of treatment
9. Recent (within 4 weeks) episode of infection requiring systemic antibiotics
10. Any medical condition that would be predicted to be exacerbated by therapy or that would limit study participation
11. Any medical condition requiring or likely to require chronic systemic administration of corticosteroids or other immunosuppressive medications during the course of this study
12. Human immunodeficiency virus (HIV) or Hepatitis B Virus (HBV) co-infection
13. Hepatocellular carcinoma (HCC) (Patients with HCC who are listed for liver transplantation may be included.)
14. Other significant chronic liver disease diagnosis
15. Evidence of decompensated liver disease
16. Solid organ transplant recipient (Patients who have a history of renal transplant, and have experienced kidney graft loss, and are not on immunosuppression may be included.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who achieve sustained virologic response | Up to 12 weeks after discontinuation of all therapy
  Primary efficacy is the proportion of patients who achieve sustained virologic response at week 12 after discontinuation of all therapy (SVR12).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth C Verna, MD, MS, Principal Investigator — Columbia University